CLINICAL TRIAL: NCT06429657
Title: Ketamine for Sedation in Severe Traumatic Brain Injury
Acronym: Ketamine
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: administrative hold at current open site and awaiting site startup at additional participating sites
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.2024.025
Record Dates: First submitted 2024-04-16; First posted 2024-05-28 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Severe Traumatic Brain Injury; Intracranial Hypertension; Intracranial Hemorrhage, Hypertensive
Keywords: TBI; Severe TBI; Traumatic Brain Injury; Sedation; Ketamine
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension; Intracranial Hemorrhage, Hypertensive | interventions — Ketamine; Propofol; Fentanyl; Dexmedetomidine; Morphine; Hydromorphone; Midazolam; Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine with propofol (Experimental): Propofol at a rate of 300 mcg/kg/hr (5 mcg/kg/min) with the addition of ketamine at a rate of 1000-5000 mcg/kg/hr (16.67 - 83.33 mcg/kg/min) (using weight at time of admission) with an additional 2 mg/kg (2000 mcg/kg) bolus of ketamine
  Interventions: Drug: Ketamine with propofol
- SOC propofol, fentanyl, dexmedetomidine, morphine, hydromorphone, midazolam, or lorazepam (Active Comparator): Standard of Care analgosedation of choice using propofol, fentanyl, dexmedetomidine, morphine, hydromorphone, midazolam, or lorazepam.
  Interventions: Other: Standard of Care propofol, fentanyl, dexmedetomidine, morphine, hydromorphone, midazolam, or lorazepam

INTERVENTIONS:
Drug: Ketamine with propofol — Propofol at a rate of 300 mcg/kg/hr (5 mcg/kg/min) with the addition of ketamine at a rate of 1000-5000 mcg/kg/hr (16.67 - 83.33 mcg/kg/min) (using weight at time of admission) with an additional 2 mg/kg (2000 mcg/kg) bolus of ketamine
  Arms: Ketamine with propofol
Other: Standard of Care propofol, fentanyl, dexmedetomidine, morphine, hydromorphone, midazolam, or lorazepam — Standard of Care analgosedation of choice using propofol, fentanyl, dexmedetomidine, morphine, hydromorphone, midazolam, or lorazepam administered according to the institutional SOC guidelines.
  Arms: SOC propofol, fentanyl, dexmedetomidine, morphine, hydromorphone, midazolam, or lorazepam

SUMMARY:
This protocol is for an open-label randomized trial evaluating the safety of using ketamine in combination with propofol for sedation versus the standard of care analgosedation in patients admitted to the intensive care unit with severe traumatic brain injury.

DETAILED DESCRIPTION:
Patients meeting eligibility criteria and consent having been obtained by LAR will undergo randomization to either the ketamine with propofol intervention arm or the standard of care control arm.

Patients enrolled in the intervention arm will receive propofol at a rate of 300 mcg/kg/hr (5 mcg/kg/min) with the addition of ketamine at a rate of 1000-5000 mcg/kg/hr (16.67 - 83.33 mcg/kg/min) (using weight at time of admission) with an additional 2 mg/kg (2000 mcg/kg) bolus of ketamine, for sustained ICP elevations over 22mHg for greater than 5 minutes not attributed to other causes (coughing etc.). In the control arm, patients will receive their institutional analgosedation protocol. The sedation protocols will be continued until removal of intracranial pressure monitoring.

This study will take place during the participant's hospital care. The clinical team will administer treatment using standard practices, including all safety precautions available. Side effects will be monitored closely and may decide to discontinue the subject's participation in the study should the subject's health or safety are at risk.

The research team will performed one outpatient follow-up after study intervention ends.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years of age
* Severe traumatic brain injury (TBI), with a Glasgow Coma Scale (GCS) ≤ 8, requiring intracranial monitoring
* Placement of intracranial pressure monitor
* Receiving treatment in an intensive care unit (ICU)

Exclusion Criteria:

* Significant cardiovascular disease with recent coronary intervention
* Pregnancy
* Prisoners
* Known allergy to ketamine or propofol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of ICP elevations greater than 22 mmHg for greater than 5 minutes | During the maximum 5-day course of study intervention, while patient is sedated and has intracranial pressure monitor in place in the ICU setting
  ICP elevations > 22 mmHg for greater than 5 minutes.
Mean ICP | During the maximum 5-day course of study intervention.
  Mean ICP

SECONDARY OUTCOMES:
Total time spent with intracranial pressure (ICP) >22 mmHg | During the maximum 5-day course of study intervention.
  Total time spent with ICP >22 mmHg (in minutes).
Mean Cerebral Perfusion Pressure (CPP) | During the maximum 5-day course of study intervention.
  Mean CPP (in minutes).
Total time spent with CPP <60 mmHg | During the maximum 5-day course of study intervention.
  Total time spent with CPP <60 mmHg (in minutes).
Total number of events where CPP <60 mmHg for greater than 5 minutes | During the maximum 5-day course of study intervention.
  Total number of events where CPP <60 mmHg (in minutes) for greater than 5 minutes.
Vasopressor dependency index (VDI) | During the maximum 5-day course of study intervention.
  Relationship between vasopressor infusion dose and mean arterial blood pressure. VDI= (dobutamine dose × 1) + (dopamine dose × 1) + (norepinephrine dose × 100) + (vasopressin × 100) + (epinephrine × 100))/MAP indicating the relationship of high VDI and poor outcome.
Incidence of seizures | During the maximum 5-day course of study intervention.
  Incidence of seizures (as documented by EEG).
Incidence of cardiac arrhythmias | During the maximum 5-day course of study intervention.
  Incidence of cardiac arrhythmias (other than sinus tachycardia).
Mean heart rate | During the maximum 5-day course of study intervention.
  Mean heart rate (HR).
Incidence of post-traumatic stress disorder (PTSD) in outpatient setting | Outpatient follow-up six months after intervention.
  Incidence of PTSD at 6-month outpatient follow-up.
Glasgow Coma Outcome Scale extended (GOSE-TBI) scores | Outpatient follow-up six months after intervention.
  GOSE-TBI assessment resulting in subjective measure of 0-8 regarding recovery after injury with higher score indicating greatest recovery to pre-injury life, will be conducted at 6-month outpatient follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Dengler, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iaccarino C, Carretta A, Nicolosi F, Morselli C. Epidemiology of severe traumatic brain injury. J Neurosurg Sci. 2018 Oct;62(5):535-541. doi: 10.23736/S0390-5616.18.04532-0. PMID 30182649
- [Background] Agrawal D, Raghavendran K, Schaubel DE, Mishra MC, Rajajee V. A Propensity Score Analysis of the Impact of Invasive Intracranial Pressure Monitoring on Outcomes after Severe Traumatic Brain Injury. J Neurotrauma. 2016 May 1;33(9):853-8. doi: 10.1089/neu.2015.4015. Epub 2015 Oct 8. PMID 26414629
- [Background] Butcher I, Maas AI, Lu J, Marmarou A, Murray GD, Mushkudiani NA, McHugh GS, Steyerberg EW. Prognostic value of admission blood pressure in traumatic brain injury: results from the IMPACT study. J Neurotrauma. 2007 Feb;24(2):294-302. doi: 10.1089/neu.2006.0032. PMID 17375994
- [Background] McHugh GS, Engel DC, Butcher I, Steyerberg EW, Lu J, Mushkudiani N, Hernandez AV, Marmarou A, Maas AI, Murray GD. Prognostic value of secondary insults in traumatic brain injury: results from the IMPACT study. J Neurotrauma. 2007 Feb;24(2):287-93. doi: 10.1089/neu.2006.0031. PMID 17375993
- [Background] Murray GD, Butcher I, McHugh GS, Lu J, Mushkudiani NA, Maas AI, Marmarou A, Steyerberg EW. Multivariable prognostic analysis in traumatic brain injury: results from the IMPACT study. J Neurotrauma. 2007 Feb;24(2):329-37. doi: 10.1089/neu.2006.0035. PMID 17375997
- [Background] Petkus V, Preiksaitis A, Chaleckas E, Chomskis R, Zubaviciute E, Vosylius S, Rocka S, Rastenyte D, Aries MJ, Ragauskas A, Neumann JO. Optimal Cerebral Perfusion Pressure: Targeted Treatment for Severe Traumatic Brain Injury. J Neurotrauma. 2020 Jan 15;37(2):389-396. doi: 10.1089/neu.2019.6551. Epub 2019 Nov 13. PMID 31583962
- [Background] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000
- [Background] Cooper DJ, Rosenfeld JV, Murray L, Arabi YM, Davies AR, D'Urso P, Kossmann T, Ponsford J, Seppelt I, Reilly P, Wolfe R; DECRA Trial Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Decompressive craniectomy in diffuse traumatic brain injury. N Engl J Med. 2011 Apr 21;364(16):1493-502. doi: 10.1056/NEJMoa1102077. Epub 2011 Mar 25. PMID 21434843
- [Background] Hawryluk GWJ, Aguilera S, Buki A, Bulger E, Citerio G, Cooper DJ, Arrastia RD, Diringer M, Figaji A, Gao G, Geocadin R, Ghajar J, Harris O, Hoffer A, Hutchinson P, Joseph M, Kitagawa R, Manley G, Mayer S, Menon DK, Meyfroidt G, Michael DB, Oddo M, Okonkwo D, Patel M, Robertson C, Rosenfeld JV, Rubiano AM, Sahuquillo J, Servadei F, Shutter L, Stein D, Stocchetti N, Taccone FS, Timmons S, Tsai E, Ullman JS, Vespa P, Videtta W, Wright DW, Zammit C, Chesnut RM. A management algorithm for patients with intracranial pressure monitoring: the Seattle International Severe Traumatic Brain Injury Consensus Conference (SIBICC). Intensive Care Med. 2019 Dec;45(12):1783-1794. doi: 10.1007/s00134-019-05805-9. Epub 2019 Oct 28. PMID 31659383
- [Background] Hutchinson PJ, Kolias AG, Timofeev IS, Corteen EA, Czosnyka M, Timothy J, Anderson I, Bulters DO, Belli A, Eynon CA, Wadley J, Mendelow AD, Mitchell PM, Wilson MH, Critchley G, Sahuquillo J, Unterberg A, Servadei F, Teasdale GM, Pickard JD, Menon DK, Murray GD, Kirkpatrick PJ; RESCUEicp Trial Collaborators. Trial of Decompressive Craniectomy for Traumatic Intracranial Hypertension. N Engl J Med. 2016 Sep 22;375(12):1119-30. doi: 10.1056/NEJMoa1605215. Epub 2016 Sep 7. PMID 27602507
- [Background] Oddo M, Crippa IA, Mehta S, Menon D, Payen JF, Taccone FS, Citerio G. Optimizing sedation in patients with acute brain injury. Crit Care. 2016 May 5;20(1):128. doi: 10.1186/s13054-016-1294-5. PMID 27145814
- [Background] Stein DM, Hu PF, Brenner M, Sheth KN, Liu KH, Xiong W, Aarabi B, Scalea TM. Brief episodes of intracranial hypertension and cerebral hypoperfusion are associated with poor functional outcome after severe traumatic brain injury. J Trauma. 2011 Aug;71(2):364-73; discussion 373-4. doi: 10.1097/TA.0b013e31822820da. PMID 21825940
- [Background] Gardner AE, Dannemiller FJ, Dean D. Intracranial cerebrospinal fluid pressure in man during ketamine anesthesia. Anesth Analg. 1972 Sep-Oct;51(5):741-5. No abstract available. PMID 4672167
- [Background] Gibbs JM. The effect of intravenous ketamine on cerebrospinal fluid pressure. Br J Anaesth. 1972 Dec;44(12):1298-302. doi: 10.1093/bja/44.12.1298. No abstract available. PMID 4650346
- [Background] Green SM, Andolfatto G, Krauss BS. Ketamine and intracranial pressure: no contraindication except hydrocephalus. Ann Emerg Med. 2015 Jan;65(1):52-4. doi: 10.1016/j.annemergmed.2014.08.025. Epub 2014 Sep 20. No abstract available. PMID 25245275
- [Background] Gregers MCT, Mikkelsen S, Lindvig KP, Brochner AC. Ketamine as an Anesthetic for Patients with Acute Brain Injury: A Systematic Review. Neurocrit Care. 2020 Aug;33(1):273-282. doi: 10.1007/s12028-020-00975-7. PMID 32328972
- [Background] Laws JC, Vance EH, Betters KA, Anderson JJ, Fleishman S, Bonfield CM, Wellons JC 3rd, Xu M, Slaughter JC, Giuse DA, Patel N, Jordan LC, Wolf MS. Acute Effects of Ketamine on Intracranial Pressure in Children With Severe Traumatic Brain Injury. Crit Care Med. 2023 May 1;51(5):563-572. doi: 10.1097/CCM.0000000000005806. Epub 2023 Feb 21. PMID 36825892
- [Background] Dengler BA, Karam O, Barthol CA, Chance A, Snider LE, Mundy CM, Bounajem MT, Johnson WC, Maita MM, Mendez-Gomez PM, Seifi A, Hafeez S. Ketamine Boluses Are Associated with a Reduction in Intracranial Pressure and an Increase in Cerebral Perfusion Pressure: A Retrospective Observational Study of Patients with Severe Traumatic Brain Injury. Crit Care Res Pract. 2022 May 21;2022:3834165. doi: 10.1155/2022/3834165. eCollection 2022. PMID 35637760
- [Background] Bebarta VS, Mora AG, Bebarta EK, Reeves LK, Maddry JK, Schauer SG, Lairet JR. Prehospital Use of Ketamine in the Combat Setting: A Sub-Analysis of Patients With Head Injuries Evaluated in the Prospective Life Saving Intervention Study. Mil Med. 2020 Jan 7;185(Suppl 1):136-142. doi: 10.1093/milmed/usz302. PMID 32074369
- [Background] Hill GJ, April MD, Maddry JK, Schauer SG. Prehospital ketamine administration to pediatric trauma patients with head injuries in combat theaters. Am J Emerg Med. 2019 Aug;37(8):1455-1459. doi: 10.1016/j.ajem.2018.10.046. Epub 2018 Oct 22. PMID 30528051
- [Background] Maheswari N, Panda NB, Mahajan S, Luthra A, Pattnaik S, Bhatia N, Karthigeyan M, Kaloria N, Chauhan R, Soni S, Jangra K, Bhagat H. Ketofol as an Anesthetic Agent in Patients With Isolated Moderate to Severe Traumatic Brain Injury: A Prospective, Randomized Double-blind Controlled Trial. J Neurosurg Anesthesiol. 2023 Jan 1;35(1):49-55. doi: 10.1097/ANA.0000000000000774. Epub 2021 May 13. PMID 36745167
- [Background] Dewan MC, Rattani A, Gupta S, Baticulon RE, Hung YC, Punchak M, Agrawal A, Adeleye AO, Shrime MG, Rubiano AM, Rosenfeld JV, Park KB. Estimating the global incidence of traumatic brain injury. J Neurosurg. 2018 Apr 27;130(4):1080-1097. doi: 10.3171/2017.10.JNS17352. Print 2019 Apr 1. PMID 29701556
- [Background] Stein SC, Georgoff P, Meghan S, Mizra K, Sonnad SS. 150 years of treating severe traumatic brain injury: a systematic review of progress in mortality. J Neurotrauma. 2010 Jul;27(7):1343-53. doi: 10.1089/neu.2009.1206. PMID 20392140
- [Background] Mangat HS, Wu X, Gerber LM, Shabani HK, Lazaro A, Leidinger A, Santos MM, McClelland PH, Schenck H, Joackim P, Ngerageza JG, Schmidt F, Stieg PE, Hartl R. Severe traumatic brain injury management in Tanzania: analysis of a prospective cohort. J Neurosurg. 2021 Jan 22;135(4):1190-1202. doi: 10.3171/2020.8.JNS201243. Print 2021 Oct 1. PMID 33482641
- [Background] Howard JT, Stewart IJ, Amuan M, Janak JC, Pugh MJ. Association of Traumatic Brain Injury With Mortality Among Military Veterans Serving After September 11, 2001. JAMA Netw Open. 2022 Feb 1;5(2):e2148150. doi: 10.1001/jamanetworkopen.2021.48150. PMID 35147684
- [Background] Rutherford GW, Wlodarczyk RC. Distant sequelae of traumatic brain injury: premature mortality and intracranial neoplasms. J Head Trauma Rehabil. 2009 Nov-Dec;24(6):468-74. doi: 10.1097/HTR.0b013e3181c133d2. PMID 19940680
- [Background] Kang HK, Bullman TA. Mortality among U.S. veterans of the Persian Gulf War. N Engl J Med. 1996 Nov 14;335(20):1498-504. doi: 10.1056/NEJM199611143352006. PMID 8890102
- [Background] Bollinger MJ, Schmidt S, Pugh JA, Parsons HM, Copeland LA, Pugh MJ. Erosion of the healthy soldier effect in veterans of US military service in Iraq and Afghanistan. Popul Health Metr. 2015 Mar 18;13:8. doi: 10.1186/s12963-015-0040-6. eCollection 2015. PMID 25798075
- [Background] Dismuke CE, Walker RJ, Egede LE. Utilization and Cost of Health Services in Individuals With Traumatic Brain Injury. Glob J Health Sci. 2015 Apr 19;7(6):156-69. doi: 10.5539/gjhs.v7n6p156. PMID 26153156
- [Background] Bullock MR, Chesnut R, Ghajar J, Gordon D, Hartl R, Newell DW, Servadei F, Walters BC, Wilberger JE; Surgical Management of Traumatic Brain Injury Author Group. Surgical management of acute epidural hematomas. Neurosurgery. 2006 Mar;58(3 Suppl):S7-15; discussion Si-iv. PMID 16710967
- [Background] Bullock MR, Chesnut R, Ghajar J, Gordon D, Hartl R, Newell DW, Servadei F, Walters BC, Wilberger JE; Surgical Management of Traumatic Brain Injury Author Group. Surgical management of acute subdural hematomas. Neurosurgery. 2006 Mar;58(3 Suppl):S16-24; discussion Si-iv. PMID 16710968
- [Background] Bullock MR, Chesnut R, Ghajar J, Gordon D, Hartl R, Newell DW, Servadei F, Walters BC, Wilberger J; Surgical Management of Traumatic Brain Injury Author Group. Surgical management of traumatic parenchymal lesions. Neurosurgery. 2006 Mar;58(3 Suppl):S25-46; discussion Si-iv. doi: 10.1227/01.NEU.0000210365.36914.E3. PMID 16540746
- [Background] Donnelly J, Czosnyka M, Adams H, Cardim D, Kolias AG, Zeiler FA, Lavinio A, Aries M, Robba C, Smielewski P, Hutchinson PJA, Menon DK, Pickard JD, Budohoski KP. Twenty-Five Years of Intracranial Pressure Monitoring After Severe Traumatic Brain Injury: A Retrospective, Single-Center Analysis. Neurosurgery. 2019 Jul 1;85(1):E75-E82. doi: 10.1093/neuros/nyy468. PMID 30476233
- [Background] Farahvar A, Gerber LM, Chiu YL, Carney N, Hartl R, Ghajar J. Increased mortality in patients with severe traumatic brain injury treated without intracranial pressure monitoring. J Neurosurg. 2012 Oct;117(4):729-34. doi: 10.3171/2012.7.JNS111816. Epub 2012 Aug 17. PMID 22900846
- [Background] Badri S, Chen J, Barber J, Temkin NR, Dikmen SS, Chesnut RM, Deem S, Yanez ND, Treggiari MM. Mortality and long-term functional outcome associated with intracranial pressure after traumatic brain injury. Intensive Care Med. 2012 Nov;38(11):1800-9. doi: 10.1007/s00134-012-2655-4. Epub 2012 Aug 3. PMID 23011528
- [Background] Marshall LF, Smith RW, Shapiro HM. The outcome with aggressive treatment in severe head injuries. Part I: the significance of intracranial pressure monitoring. J Neurosurg. 1979 Jan;50(1):20-5. doi: 10.3171/jns.1979.50.1.0020. No abstract available. PMID 758374
- [Background] Lowell HM, Bloor BM. The effect of increased intracranial pressure on cerebrovascular hemodynamics. J Neurosurg. 1971 Jun;34(6):760-9. doi: 10.3171/jns.1971.34.6.0760. No abstract available. PMID 4997951
- [Background] Akerlund CA, Donnelly J, Zeiler FA, Helbok R, Holst A, Cabeleira M, Guiza F, Meyfroidt G, Czosnyka M, Smielewski P, Stocchetti N, Ercole A, Nelson DW; CENTER-TBI High Resolution ICU Sub-Study Participants and Investigators. Impact of duration and magnitude of raised intracranial pressure on outcome after severe traumatic brain injury: A CENTER-TBI high-resolution group study. PLoS One. 2020 Dec 14;15(12):e0243427. doi: 10.1371/journal.pone.0243427. eCollection 2020. PMID 33315872
- [Background] Sheth KN, Stein DM, Aarabi B, Hu P, Kufera JA, Scalea TM, Hanley DF. Intracranial pressure dose and outcome in traumatic brain injury. Neurocrit Care. 2013 Feb;18(1):26-32. doi: 10.1007/s12028-012-9780-3. PMID 23055087
- [Background] Wolf S, Mielke D, Barner C, Malinova V, Kerz T, Wostrack M, Czorlich P, Salih F, Engel DC, Ehlert A, Staykov D, Alturki AY, Sure U, Bardutzky J, Schroeder HWS, Schurer L, Beck J, Juratli TA, Fritsch M, Lemcke J, Pohrt A, Meyer B, Schwab S, Rohde V, Vajkoczy P; EARLYDRAIN Study Group. Effectiveness of Lumbar Cerebrospinal Fluid Drain Among Patients With Aneurysmal Subarachnoid Hemorrhage: A Randomized Clinical Trial. JAMA Neurol. 2023 Aug 1;80(8):833-842. doi: 10.1001/jamaneurol.2023.1792. PMID 37330974
- [Background] Cooper DJ, Nichol AD, Bailey M, Bernard S, Cameron PA, Pili-Floury S, Forbes A, Gantner D, Higgins AM, Huet O, Kasza J, Murray L, Newby L, Presneill JJ, Rashford S, Rosenfeld JV, Stephenson M, Vallance S, Varma D, Webb SAR, Trapani T, McArthur C; POLAR Trial Investigators and the ANZICS Clinical Trials Group. Effect of Early Sustained Prophylactic Hypothermia on Neurologic Outcomes Among Patients With Severe Traumatic Brain Injury: The POLAR Randomized Clinical Trial. JAMA. 2018 Dec 4;320(21):2211-2220. doi: 10.1001/jama.2018.17075. PMID 30357266
- [Background] Roquilly A, Moyer JD, Huet O, Lasocki S, Cohen B, Dahyot-Fizelier C, Chalard K, Seguin P, Jeantrelle C, Vermeersch V, Gaillard T, Cinotti R, Demeure Dit Latte D, Mahe PJ, Vourc'h M, Martin FP, Chopin A, Lerebourg C, Flet L, Chiffoleau A, Feuillet F, Asehnoune K; Atlanrea Study Group and the Societe Francaise d'Anesthesie Reanimation (SFAR) Research Network. Effect of Continuous Infusion of Hypertonic Saline vs Standard Care on 6-Month Neurological Outcomes in Patients With Traumatic Brain Injury: The COBI Randomized Clinical Trial. JAMA. 2021 May 25;325(20):2056-2066. doi: 10.1001/jama.2021.5561. PMID 34032829
- [Background] Skolnick BE, Maas AI, Narayan RK, van der Hoop RG, MacAllister T, Ward JD, Nelson NR, Stocchetti N; SYNAPSE Trial Investigators. A clinical trial of progesterone for severe traumatic brain injury. N Engl J Med. 2014 Dec 25;371(26):2467-76. doi: 10.1056/NEJMoa1411090. Epub 2014 Dec 10. PMID 25493978
- [Background] CRASH-3 trial collaborators. Effects of tranexamic acid on death, disability, vascular occlusive events and other morbidities in patients with acute traumatic brain injury (CRASH-3): a randomised, placebo-controlled trial. Lancet. 2019 Nov 9;394(10210):1713-1723. doi: 10.1016/S0140-6736(19)32233-0. Epub 2019 Oct 14. PMID 31623894
- [Background] Bourgoin A, Albanese J, Wereszczynski N, Charbit M, Vialet R, Martin C. Safety of sedation with ketamine in severe head injury patients: comparison with sufentanil. Crit Care Med. 2003 Mar;31(3):711-7. doi: 10.1097/01.CCM.0000044505.24727.16. PMID 12626974
- [Background] Bourgoin A, Leone M, Delmas A, Garnier F, Albanese J, Martin C. Increasing mean arterial pressure in patients with septic shock: effects on oxygen variables and renal function. Crit Care Med. 2005 Apr;33(4):780-6. doi: 10.1097/01.ccm.0000157788.20591.23. PMID 15818105
- [Background] Kolenda H, Gremmelt A, Rading S, Braun U, Markakis E. Ketamine for analgosedative therapy in intensive care treatment of head-injured patients. Acta Neurochir (Wien). 1996;138(10):1193-9. doi: 10.1007/BF01809750. PMID 8955439
- [Background] Schmittner MD, Vajkoczy SL, Horn P, Bertsch T, Quintel M, Vajkoczy P, Muench E. Effects of fentanyl and S(+)-ketamine on cerebral hemodynamics, gastrointestinal motility, and need of vasopressors in patients with intracranial pathologies: a pilot study. J Neurosurg Anesthesiol. 2007 Oct;19(4):257-62. doi: 10.1097/ANA.0b013e31811f3feb. PMID 17893578
- [Background] Sakpal TV. Sample size estimation in clinical trial. Perspect Clin Res. 2010 Apr;1(2):67-9. PMID 21829786
- [Background] Military Health System and Defense Health Agency. DOD TBI Worldwide Numbers: Traumatic Brain Injury Center of Excellence; 2022 [Available from: https://health.mil/Military-Health-Topics/Centers-of-Excellence/Traumatic-Brain-Injury-Center-of-Excellence/DOD-TBI-Worldwide-NumbersTraumaticBrain].
- [Background] Michalczyk, Lukasz, and Lukasz Kaczmarek.
- [Background] Chan, Kai En, et al.